CLINICAL TRIAL: NCT00911495
Title: Phase 1/Phase 2 Study of the Safety, Pharmacokinetics, and Microvascular Effect of Titrating Doses of Intravenous GMI-1070, a Pan-Selectin Inhibitor, in Adults With Sickle Cell Disease
Brief Title: Study of Intravenous GMI-1070 in Adults With Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMI-1070-103
Record Dates: First submitted 2009-05-27; First posted 2009-06-02 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — rivipansel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GMI-1070 (Experimental)
  Interventions: Drug: GMI-1070

INTERVENTIONS:
Drug: GMI-1070 — Intravenous GMI-1070 given as two doses over the course of one day

SUMMARY:
This Phase 1/Phase 2 study will evaluate GMI-1070, a pan-selectin inhibitor, in adults with stable sickle cell disease. The study will assess safety, pharmacokinetics, and microvascular effects of intravenous GMI-1070 in the outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years
* Established diagnosis of SCD-SS or SCD-SB0-thal
* At medical baseline, with no evidence of worsening of disease over the last 3 months
* Available and agree to return for follow-up visits for the full duration of the study
* Able to cooperate with study procedures
* Documented and observed written informed consent

Exclusion Criteria:

* Vaso-occlusive crisis
* Recent major surgery, hospitalization, infection, significant bleeding, cerebrovascular accident or seizure, or transfusion
* Currently receiving, or has received within the previous 4 weeks, any other investigational agent
* Pregnant or lactating female; or female of childbearing age unable or unwilling to comply with birth control or abstinence during the course of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Thackray, MD, Study Director — GlycoMimetics Incorporated
Locations (3):
- United States (3):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - University of California at Davis, CCRC, Sacramento, California
  - Duke Comprehensive Sickle Cell Center, Durham, North Carolina

REFERENCES:
- [Derived] Wun T, Styles L, DeCastro L, Telen MJ, Kuypers F, Cheung A, Kramer W, Flanner H, Rhee S, Magnani JL, Thackray H. Phase 1 study of the E-selectin inhibitor GMI 1070 in patients with sickle cell anemia. PLoS One. 2014 Jul 2;9(7):e101301. doi: 10.1371/journal.pone.0101301. eCollection 2014. PMID 24988449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 28 May 2009; last subject completed 6 July 2010.
Groups:
- GMI-1070: GMI-1070 administered IV at 20 mg/kg loading dose, followed by a single dose of 10 mg/kg in the evening
Period: Overall Study
Arm/Group | GMI-1070
Started | 15
Completed | 14
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | GMI-1070
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 28 [19 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by the Number of Participants With Adverse Events
Time Frame: 28 days
Population: All enrolled subjects were analyzed for safety.
Measure: Number; unit: participants
Arm/Group | GMI-1070
Number analyzed (Participants) | 15
participants | 9

2. Secondary Outcome: Total Plasma Clearance
Time Frame: 48 hours
Population: All subjects were analyzed for pharmacokinetics; one subject of the 15 enrolled was lost to follow-up.
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | GMI-1070
Number analyzed (Participants) | 14
mL/h/kg | 19.6 (6.42)

3. Other Pre Specified Outcome: Blood Flow and Biomarkers of Adhesion
Description: As an exploratory outcome mean change in microvascular blood flow from baseline to each time point was measured. Microvascular blood flow was also measured as microFI, perfused vessel density, and RBC velocity.
Time Frame: 48 hours
Reporting Status: Not Posted

4. Secondary Outcome: Volume of the Central Compartment
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | GMI-1070
Number analyzed (Participants) | 14
mL/kg | 120 (30.7)

5. Secondary Outcome: Intercompartmental Clearance
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | GMI-1070
Number analyzed (Participants) | 14
mL/h/kg | 31.6 (17.2)

6. Secondary Outcome: Volume of the Peripheral Compartment
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | GMI-1070
Number analyzed (Participants) | 14
mL/kg | 64.2 (19.6)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | GMI-1070
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 9/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GMI-1070 (N=15)
Headache (Nervous system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
sickle cell anemia with crisis (Congenital, familial and genetic disorders) | 2
vomiting (Gastrointestinal disorders) | 1
infusion site pain (General disorders) | 1
hypokalemia (Metabolism and nutrition disorders) | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less